CLINICAL TRIAL: NCT06528665
Title: A Pharmacokinetic, Safety and Tolerability Formulation Screening Comparing Corplex Ozanimod TDS to Oral Ozanimod Capsules in Healthy Adults Subjects
Brief Title: Determine PK Profiles of Ozanimod and Its' Major Metabolites in Healthy Subjects
Status: Recruiting | Type: Observational
Sponsor: Corium Innovations, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OZ101A
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis; Ulcerative Colitis
Keywords: Ozanimod; Transdermal Delivery system; Pharmacokinetics
MeSH Terms: conditions — Multiple Sclerosis; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- 4 groups subjects will be recruited. Each group will be composed of 6 subjects, sex ratio 1:1: Group1, 2,3 will be administered with 3 different patches (TDS) once for a week, respectively; Group 4 will be oral administered with one capsule (0.92 mg) only.
  Interventions: Drug: ZEPOSIA® indicated for the treatment of: Relapsing forms of multiple sclerosis, and active ulcerative colitis in adults

INTERVENTIONS:
Drug: ZEPOSIA® indicated for the treatment of: Relapsing forms of multiple sclerosis, and active ulcerative colitis in adults — ZEPOSIA®
  * Titration is required for treatment initiation.
  * The recommended maintenance dosage is 0.92 mg orally once daily.
  * If a dose is missed within the first 2 weeks of treatment, reinitiate with the titration regimen. If a dose is missed after the first 2 weeks of treatment, continue treatment as planned.

SUMMARY:
The goal of this clinical trial is to learn how Ozanimod drug can be administered to the healthy subjects via transdermal delivery system (TDS, patch) to achieve better drug absorption and delivery than via oral capsules (Zeposia). Researchers will compare two administered routes of Ozanimod TDS and oral Zeposia in drug pharmacokinetics, tolerability and safety. Participants will either take one capsule only or wear a patch on his/her arm for 7 days, and blood samples will be collected to measure drug concentrations and local skin reactions will be also observed.

DETAILED DESCRIPTION:
This is a single-dose, single-center, open-label, randomized, parallel relative bioavailability study (4 treatments and 1 period) of 3 test products of a Transdermal Delivery System of Ozanimod (Corplex Ozanimod TDS) with the Reference Listed Drug (Zeposia Capsule 0.92 mg), recruiting around 24 healthy (male: female = 1:1) subjects under fasting conditions.

The following goals will be procured through this study:

1. To determine the pharmacokinetic profiles of Ozanimod and its' major metabolites (CC112273 and CC1084037) from the Corplex Ozanimod TDS (OZ-TDS 1, OZ-TDS 2 and OZ-TDS 3 manufactured by Corium Innovations, Inc.) (Test Product 1, Test Product 2 and Test Product 3) and the comparator (Zeposia Capsule 0.92 mg manufactured by Bristol Myers Squibb) (Reference Product) in healthy subjects;
2. To compare the relative bioavailability between the Corplex Ozanimod TDS and the oral capsules in healthy subjects;
3. To compare three formulations of the Corplex Ozanimod TDS in healthy subjects;
4. To determine the safety and tolerability of the Corplex Ozanimod TDS vs the oral capsules in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age between 18 to 55 years old.
2. Subject body weight ≤ 120 kg, with a BMI within 18-30 kg/m2.
3. Subject is able to complete the clinical study including the follow-up.
4. Subject is capable of providing written informed consent.

Exclusion Criteria:

1. Breastfeeding female.
2. Pregnancy test positive female.
3. At rest systolic blood pressure outside 90-140 mmHg or diastolic blood pressure outside 50-90 mmHg.
4. At rest sinus bradycardia defined as symptomatic heart rate < 50 bpm, or asymptomatic heart rate < 45 bpm; and sinus tachycardia defined as heart rate > 100 bpm.
5. Clinically significant ECG abnormalities or Participant with history or presence of second-degree atrioventricular (AV) block Type II or third-degree AV block or sick sinus syndrome unless the patient has a functioning pacemaker.
6. QTc > 450 ms for male and > 460 ms for female.
7. A history of allergies, or any significant adverse reactions, to any medications, unless the clinician considers that they are not clinically significant.
8. Clinically significant medical history of eyes, ears, nose, throat, respiratory, cardiovascular, gastrointestinal, genitourinary, neurological, haematopoietic, lymphatic, endocrine, metabolic, dermatological, musculoskeletal, psychological, family history or surgical history.
9. Family history of sudden cardiac death.
10. Clinically significant physical examination finding.
11. Clinically significant laboratory abnormalities.
12. Haemoglobin < 12.0 g/dL for male and < 11.0 g/dL for female at screening.
13. Total bilirubin > 1.25 x upper limit of normal (unless it is an isolated elevation where the direct bilirubin is ≤ 35% of total), ALT/AST > 1.5 x upper limit of normal, or CK > 2 x upper limit of normal.
14. Hepatitis B, Hepatitis C or HIV positive.
15. Urine DOA test positive.
16. Breath alcohol test positive.
17. Any use of tobacco product(s) 30 days prior to study recruitment.
18. A history of drug or substance abuse, including alcohol (≥ 14 units per week) within 6 months before consent taking (1 unit of alcohol equals approximately ½ pint [285 mL] of beer, 1 glass [125 mL] of wine, or 1 shot [25 mL] of spirit).
19. Unable to refrain from taking any medications (including herbal remedies) within 7 days before dosing, with the exception of birth control medications and other medications deemed acceptable by the Investigator.
20. Clinically significant illness or injury or hospitalisation for any reason within 28 days before consent-taking.
21. Unable to refrain or has participation in other clinical study involving a marketed or investigational drug within 28 days or 10 half-lives of the drug before dosing, whichever is longer.
22. Unable to refrain or has donation of > 500 mL of plasma within 14 days before dosing; or donation or loss of whole blood (excluding the amount of blood collected during screening) before dosing as follows:

    * 50-300 mL within 28 days,
    * 301-500 mL within 42 days, or
    * > 500 mL within 84 days.
23. Any upper arm conditions that will disallow study drug administration or difficulty to swallow the study drug.
24. Any other medical condition or reason that, in the opinion of the Investigator or Research Physician, makes the subject unsuitable to participate in the clinical study.
25. Unable to refrain from taking any of the following systemic medications:

    Strong inhibitors of CYP3A, and all inhibitors of CYP2C8 or BCRP, (i.e., cyclosporine eltrombopag, geftinib) within 7 days or 5 half-lives, whichever is longer, prior to dosing or Strong inducers of CYP3A, and all inducers of CYP2C8 within 14 days or 5 half-lives, whichever is longer, prior to dosing, or Any known MAO inhibitors within 30 days or 5 half-lives, whichever is longer, prior to Day 1.

    Examples of MAO inhibitors include but are not limited to phenelzine, selegiline, isocarboxazid, rasagiline, tranylcypromine, pargyline, procarbazine, and furazolidone.
26. Female of childbearing potential unable to refrain from having unprotected sexual intercourse with any non-sterile male partner within 14 days before dosing; acceptable methods of contraception include:

    * double barrier (1 by each partner), and at least 1 of these barriers (condom, cervical cap, diaphragm or sponge) must contain spermicide,
    * hormonal (oral, injectable, transdermal, intravaginal or implantable),
    * intrauterine contraceptive system,
    * surgical (vasectomy or tubal ligation), or
    * sexual abstinence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological sex
Study Population: Local subjects participate in the Hospital Ampang, Malaysia
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-16 (Estimated); Study Completion 2025-04-16 (Estimated)

PRIMARY OUTCOMES:
Plasma Pharmacokinetic- AUC 0-t (Ozanimod, CC112273, CC1084037) | 15 days
  area under the concentration-time curve from time-zero to the time of the last quantifiable concentration
Plasma Pharmacokinetic- AUC 0-∞ (Ozanimod, CC112273, CC1084037) | 15 days
  area under the concentration-time curve from time-zero to infinity
Plasma Pharmacokinetic- Cmax (Ozanimod, CC112273, CC1084037) | 15 days
  Peak concentration within the dosing interval
Plasma Pharmacokinetic- Tmax (Ozanimod, CC112273, CC1084037) | 15 days
  Time to peak concentration (Cmax)
Plasma Pharmacokinetic- T 1/2 (Ozanimod, CC112273, CC1084037) | 15 days
  Terminal elimination half-life
Plasma Pharmacokinetic- MTR(Ozanimod, CC112273, CC1084037) | 15 days
  Mean residence time
Plasma Pharmacokinetic-Lambda z(λz) (Ozanimod, CC112273, CC1084037) | 15 days
  Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Damenthi Nair, MD, Principal Investigator — Hospital Ampang, 68000 Ampang, Malaysia
Locations (1):
- Hospital Ampang, Ampang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran JQ, Zhang P, Ghosh A, Liu L, Syto M, Wang X, Palmisano M. Single-Dose Pharmacokinetics of Ozanimod and its Major Active Metabolites Alone and in Combination with Gemfibrozil, Itraconazole, or Rifampin in Healthy Subjects: A Randomized, Parallel-Group, Open-Label Study. Adv Ther. 2020 Oct;37(10):4381-4395. doi: 10.1007/s12325-020-01473-0. Epub 2020 Aug 28. PMID 32857315